CLINICAL TRIAL: NCT06916221
Title: Behavioral Intervention Development Core - Long Term Memory Digital Intervention in Aging
Brief Title: BID LTM Digital Intervention in Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-43268; P30AG086635 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Long-Term Memory; Inhibitory Control; Mild Cognitive Impairment
Keywords: cognitive training; cognitive aging; memory
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Long Short Term Memory

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After recruitment, participants are randomly assigned to one of two arms, Participants and experimenters with whom they interact during the experiment are blind to treatment purpose of the randomly-assigned arm. First-level analysis of the data (baseline, post training and follow up) performed blind to the participant's arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Term Memory (Active Comparator): Multi-session cognitive intervention as a computer game that presents an adaptive spatial wayfinding challenge.
  Interventions: Behavioral: Long Term Memory
- Worder (Active Comparator): Multi-session cognitive intervention as a computer game that presents a word puzzle.
  Interventions: Behavioral: Worder

INTERVENTIONS:
Behavioral: Long Term Memory — Tablet computer game designed to stimulate environmental enrichment via an adaptive and immersive experience learning virtual neighborhoods and errands in order to complete assigned errands.
  Arms: Long Term Memory
Behavioral: Worder — Tablet computer game designed to stimulate interest in solving word puzzles, much like the Boggle game.
  Arms: Worder

SUMMARY:
Healthy aging is typically accompanied by diminished capability for learning and retrieval of high-fidelity long-term memory (LTM). The decline in these faculties is accelerated and becomes significant deficits in LTM and cognitive control functions at the level or a diagnosis of Mild Cognitive Impairment (MCI). Training with the navigation game, relative to training with control games, is expected to improve LTM performance for older adult participants.

Researchers will compare two different digital interventions to assess whether they may be helpful in improving cognitive function.

Participants will conduct study activities remotely (e.g., at-home):

1. Baseline Assessment. Complete a series of cognitive assessments and surveys.
2. Intervention. Engage in a digital intervention for up to 8 weeks.
3. Post Intervention Assessment. Complete the same cognitive assessments and surveys as the Baseline Assessment.
4. Follow-Up Assessment. Six months after the intervention ends, participants will complete the same cognitive assessments and surveys as the Baseline Assessment.

DETAILED DESCRIPTION:
Older adult participants consent and enroll in the LTM Digital Intervention, which is a randomized control trial (RCT) administered on the Neuroscape Nexus web-based research platform. Enrolled participants are randomly assigned to either of two arms that will play memory-based games.

Participants are provided by the study team with an Apple iPad 10th Generation (2024) at their home address, which will enable them to complete all study tasks at home via Nexus. All required applications will be pre-loaded on the device.

Participants will receive notifications and reminders to complete study tasks by email, through in-app reminders, or SMS. They can view their task list and progress in their personal dashboard in Nexus.

Study procedures include a series of surveys and brief tests of memory and attention as Baseline Tests, which make take up to 120 minutes and can be completed across more than one session.

Participants will engage with their assigned training application to complete 45 minutes of training, several days a week for up to 8 weeks for a total of 1000 minutes of training. Participants will be randomly assigned to one of two intervention apps, which encourage long-term memory.

Once their assigned training regimen is complete, participants will again fulfill a series of surveys and brief tests of memory and attention as Post-Training Tests, which make take up to 120 minutes and can be completed across more than one session.

Six months after completion of all Post-Training Tests, participants will be fulfill a third series of surveys and brief tests of memory and attention as Follow-Up Tests, which make take up to 120 minutes and can be completed across more than one session.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 12 years of education
* English fluency: All task instructions are presented in English language text. In order to control for sufficient and equivalent participant comprehension of the procedures and instructions, we require their self-report of fluency in English.
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing
* Medically healthy older adults, including those with below-average cognitive performance /MCI patients without dementia referred by neuropsychologists (i.e., no participant medical records will be reviewed).

Exclusion Criteria:

* Under the age of 60
* Clinical diagnosis of neurological or psychiatric disorder Clinical diagnosis of dementia or AD8 score of >4
* Visually or hearing impaired without correction to normal
* Regularly (one or more times per week) practicing an instrument within the last year
* 10 years or more of formal musical instrument training

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
MDT change in recognition memory | baseline promptly before, post-training promptly after regimen is completed, and follow up six months after post-training tests
  Psychometric test for proportion correct in memory for studied images of common objects versus paired similar lures
TOUR change in cued recall memory | baseline promptly before, post-training promptly after regimen is completed, and follow up six months after post-training tests
  Psychometric test for proportion of details correctly recalled from recent autobiographical memory

SECONDARY OUTCOMES:
Cognitive Assessment change in working memory | baseline promptly before, post-training promptly after regimen is completed, and follow up six months after post-training tests
  Psychometric test for proportion of number of correctly identified images from working memory span

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Wais, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francsico, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data to be shared includes demographic, cognitive assessments, survey, and behavioral outcomes.
Supporting Information: Study Protocol, ICF, Analytic Code